CLINICAL TRIAL: NCT04552769
Title: Abemaciclib in Metastatic or Locally Advanced Anaplastic/Undifferentiated Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Saad A Khan, ASSOCIATE PROFESSOR OF MEDICINE (ONCOLOGY), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-57905; END0023 (Other: OnCore); NCI-2020-07832 (Other: NCI Trial Identifier)
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Thyroid Cancer; Anaplastic Thyroid Cancer; Undifferentiated Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Carcinoma, Anaplastic | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Abemaciclib (Experimental): Each cycle of therapy will be 28 days long. A completed cycle will be twice daily abemaciclib. Number of Cycles: until progression or unacceptable toxicity develops
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — 200 mg orally
  Other Names: Verzenio; LY2835219; 2-pyrimidinamine, N-(5-((4-ethyl-1-piperazinyl)methyl)-2-pyridinyl)-5-fluoro-4-(4-fluoro-2-methyl-1-(1-methylethyl)-1H-benzimidazol-6-yl)

SUMMARY:
The purpose of the study is to evaluate the efficacy of treatment with abemaciclib in patients with anaplastic thyroid/undifferentiated thyroid

DETAILED DESCRIPTION:
Primary Objective The primary objective is to determine the overall response rate after treatment with abemaciclib in patients with anaplastic thyroid/undifferentiated thyroid cancer.

Secondary Objectives The secondary objectives are to describe the overall survival (OS) and progression-free survival (PFS) after treatment with abemaciclib in patients with anaplastic thyroid/undifferentiated thyroid cancer.Safety assessments of AE's will also be analysed

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of anaplastic thyroid cancer or undifferentiated thyroid cancer that does not have a known BRAF V600E positive on tissue/blood testing. BRAF V600E positive patients are eligible if they have previously received FDA approved therapy for this genetic abnormality and progressed or become intolerant.
2. Patients will be eligible if they meet either criteria:

   * Unresectable anaplastic thyroid cancer limited to the neck: Patients must have received radiation therapy or surgery to primary tumor and have subsequent evidence of anaplastic thyroid cancer (ATC).
   * Metastatic anaplastic thyroid cancer: either with entirely surgically removed cancer/metastatic only disease, or with disease in the neck not requiring radiation or surgery to the neck mass.
3. Patients with a bulky thyroid/neck mass and those in whom airway obstruction is suspected should undergo an evaluation via indirect or direct laryngoscopy to ensure patency of the trachea/airway prior to enrollment
4. Patients will not have any other curative therapeutic option, such as radiation or surgery.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
6. Have measurable disease based on RECIST 1.1
7. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived sample.
8. Be ≥ 18 years of age on day of signing informed consent.
9. Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to study treatment start. A washout period of at least 21 days is required between last chemotherapy dose and study treatment start (provided the patient did not receive radiotherapy).
10. Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and study treatment start.
11. The patient is able to swallow oral medications.
12. The patient has adequate organ function for all of the following criteria, Laboratory Value Guidance to Establish Adequate Organ Function System Laboratory Value Hematologic absolute neutrophil count (ANC)≥1.5 × 109/L Platelets≥100 × 109/L Hemoglobin≥8 g/dL Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.

    Hepatic Total bilirubin ≤1.5 × upper limit of normal(ULN) Patients with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted.

    alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤3 × ULN
13. Women of childbearing potential and all men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) while taking drug and agree to continue for 3 months after the last dose of study treatment. Women of child bearing potential and male patients for 3 months should not mother or father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
14. Patient has the ability to understand and provide signed informed consent.
15. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other procedures.

Exclusion Criteria:

1. Patients with known hypersensitivity to any of the excipients of abemaciclib
2. History of carcinomatous meningitis
3. Prior therapy with abemaciclib.
4. The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
5. Females who are pregnant or lactating.
6. The patient has active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
7. The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
8. Presence or history of a malignant disease other than thyroid cancer that has been diagnosed and/or required therapy within the past year and is undergoing active anticancer treatment. Exceptions to this exclusion include the following: completely resected basal cell and squamous cell skin cancers, and completely resected carcinoma in situ of any type.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2025-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saad A Khan, MD, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abemaciclib
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Abemaciclib
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response (OR)
Description: Overall response defined as either complete response or partial response assessed using RECIST v1.1 criteria. This measure will be reported as a number without dispersion.
  RECIST v1.1 criteria:
  Evaluation of Target Lesions Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, no appearance of new lesions.
  Evaluation of Non-Target Lesions Complete Response (CR): Disappearance of all non-target lesions Incomplete Response/Stable Disease (SD): Persistence of one or more non-target lesion(s) Progressive Disease (PD): Appearance of one or more new lesions
Time Frame: 8 (+/-4) weeks from start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Abemaciclib
Number analyzed (Participants) | 9
Participants | 0

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival defined as duration of time from start of treatment to death from any cause. This will be reported as median survival time with interquartile range
Time Frame: 3 years
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Abemaciclib
Number analyzed (Participants) | 9
days | 130 [56 to NA] — The upper bound of the inter-quartile range was not reached due to insufficient number of participants with events

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) defined as the duration of time from start of treatment to time of progression or death from any cause. This will be reported as median time with interquartile range.
Time Frame: 3 years
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Abemaciclib
Number analyzed (Participants) | 9
day | 69 [35 to 125]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Abemaciclib
All-Cause Mortality (participants affected / at risk) | 7/9
Serious Adverse Events (participants affected / at risk) | 6/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib (N=9)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tracheal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib (N=9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (13)
Nausea (Gastrointestinal disorders) | 6 (8)
Headache (Nervous system disorders) | 1 (3)
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 6 (9)
Vomitting (Gastrointestinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 3 (6)
Unilateral Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Shortness og Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Pnuemonia (Psychiatric disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Cyst NOS (Skin and subcutaneous tissue disorders) | 1 (1)
Glucose High (Endocrine disorders) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
WBC decreased (Blood and lymphatic system disorders) | 1 (4)
Foot Edema (Skin and subcutaneous tissue disorders) | 1 (1)
Creatinine Increased (Renal and urinary disorders) | 1 (1)
BUN Increased (Renal and urinary disorders) | 1 (2)
Alkaline phosphatase increased (Blood and lymphatic system disorders) | 1 (1)
ALT increased (Gastrointestinal disorders) | 1 (1)
Stomach irritated feeling of (Gastrointestinal disorders) | 1 (1)
cramps of extremities (Musculoskeletal and connective tissue disorders) | 1 (1)
UTI (Renal and urinary disorders) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1)
Hoarness of voice (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Swallowing difficult (Gastrointestinal disorders) | 1 (1)
Breathing difficult (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)
Hypermagnesemia (Blood and lymphatic system disorders) | 1 (1)
Increased creatinine clearance (Renal and urinary disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CD4 lymphocytes (Blood and lymphatic system disorders) | 1 (1)
Neutrophil count abnormal (Blood and lymphatic system disorders) | 1 (1)
Platelet count low (Blood and lymphatic system disorders) | 1 (1)
Monocyte decreased (Blood and lymphatic system disorders) | 1 (1)
RDW Increased (Blood and lymphatic system disorders) | 1 (1)
Glucose Increased (Endocrine disorders) | 1 (1)
Chlorides blood increased (Blood and lymphatic system disorders) | 1 (1)
Troponin increased (Cardiac disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Pressure Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT04552769/Prot_SAP_003.pdf